CLINICAL TRIAL: NCT03950804
Title: Transcriptome and Metabolic Analyses of CHAPLE Disease Patients With or Without Eculizumab Treatment
Brief Title: Transcriptome and Metabolic Analyses of CHAPLE Disease
Acronym: CHAPLEOMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Ahmet Ozen, M.D., Prof. Of Pediatrics, Division of Allergy and Immunology, Marmara University
Other Study IDs: 09.2018.242; ZIAAI000717-22 (NIH)
Record Dates: First submitted 2019-05-12; First posted 2019-05-15 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: CD55 - Cluster of Differentiation Antigen 55 Deficiency; Primary Intestinal Lymphangiectasis; Protein-Losing Enteropathies; Complement Regulatory Factor Defect
Keywords: Complement hyperactivation; CD55 deficiency; Complement C5; Eculizumab; Multi-OMICs Analyses; Protein losing enteropathy
MeSH Terms: conditions — Waldmann disease; Protein-Losing Enteropathies | interventions — eculizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells (PBMC) Serum Plasma Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CHAPLE patients, without eculizumab treatment: Patients with suspected CHAPLE syndrome undergo flow-cytometry based CD55 surface staining of peripheral blood samples. Those patients with loss of CD55 protein expression are diagnosed with CHAPLE syndrome. A subgroup of the CHAPLE patients describe only mild symptoms and are not treated with eculizumab, but monitored closely for any disease progression.
- Control subjects- no intervention: Healthy subjects with no history of any chronic disease. All investigational analyses are performed on both the case and the control subjects. Therefore, the same type of biological specimens collected from the case group are collected from the control group simultaneously.
- Non-CHAPLE PILs: PIL patients with intact CD55 on flow-cytometry assesment undergo genetic testing to exclude a potential missense mutation in the CD55 gene that impairs its function while retaining protein expression. Overall, patients and their parents undergo exome sequencing as trios, and examined for potential gene mutations underlying their disease. Non-CHAPLE PILs are also examined by high-throughput investigation similarly to CHAPLE patients.
- CHAPLE patients on eculizumab: Among CHAPLE patients, there is a subgroup who receive eculizumab treatment. These patients are prospectively followed and biological samples collected at baseline as well as periodically under therapy. Eculizumab (Soliris) is being provided for CHAPLE patients on an off-label basis upon approval of the physician's request of the drug by Turkish Medicines and Medical Devices Agency (TMMDA) of Turkish Ministry of Health. The dosage and interval of the drug is determined according to manufacturer's recommendations based on the weight of the patients.
  Interventions: Drug: Eculizumab Injection

INTERVENTIONS:
Drug: Eculizumab Injection — Patients receive eculizumab as deemed necessary by the primary physician
  Other Names: Soliris
  Groups: CHAPLE patients on eculizumab

SUMMARY:
CHAPLE syndrome (complement hyperactivation, angiopathic thrombosis, protein losing enteropathy) is a newly discovered genetic disorder, which is caused by deleterious mutations in the CD55 gene. Patients often suffer from chronic manifestations that may lead to life-threatening complications despite conventional treatment options.The cause of gastrointestinal protein loss is distorted lacteals in the gut, referred to as primary intestinal lymphangiectasia (PIL). There is a second group of patients with PIL with intact CD55, referred to here as "non-CHAPLE PIL". The current study aims to explore the signatures of CHAPLE and non-CHAPLE PILs, discover druggable molecular targets and identify biomarkers that can direct therapy. A subgroup of patients with CHAPLE syndrome receive treatment with a complement C5 blocker, eculizumab, on an off-label basis. This study involves serial transcriptome and metabolic profiling of biological samples under eculizumab therapy and correlates them with the clinical response. Overall, the aim of this research is to integrate clinical data and high-throughput metabolic profiling approaches to better characterize the etiology of PILs and develop novel therapeutic approaches.

DETAILED DESCRIPTION:
CHAPLE syndrome is a newly discovered genetic disorder characterized by excessive loss of proteins in the gastrointestinal tract, referred to as protein-losing enteropathy. The disease typically presents in early childhood with facial and extremity edema in relation to hypoalbuminemia, chronic diarrhea, failure to thrive and, in extreme cases, severe thromboembolic disease that can lead to premature death. Patients afflicted with this newly discovered disease have been treated with conventional medications, including inflammatory bowel disease drugs to reduce gastrointestinal inflammation, albumin and immunoglobulin replacement therapy, dietary modification, supportive measures to supplement micronutrients and vitamins, surgery to remove affected intestinal segments, among others. These interventions have often provided only partial relief, with no capacity to alter the natural course of the disease.

CHAPLE syndrome is caused by loss of a complement regulatory protein due to deleterious mutations in the CD55 gene, which results in excessive activation of the complement system. Based on the scientific observations that complement hyperactivation is the primary event that underlies disease manifestations, it was hypothesized that complement inhibition therapy can potentially reverse the pathological processes. Through a compessionate program 3 CHAPLE patients from a single family have been treated with a complement C5 blocker antibody called eculizumab, with favorable response (Kurolap et al. PMID: 28657861). While these observations confirm the primary role of complement hyper activation in PIL associated with CHAPLE syndrome, the pathogenesis of PILs not related to CD55 deficiency (non-CHAPLE PIL) remains unknown. It is hypothesized that that there may be pathogenetic intersections between CHAPLE and non-CHAPLE PILs.

Following a clinical observation that eculizumab provides a rapid clinical relief in unrelated CHAPLE patients based in Turkey similar to Kurolap et al.'s report, researchers of this study decided to evaluate the clinical outcome of eculizumab among subsequent CHAPLE patients who are placed on this therapy. In parallel, molecular investigations on biological samples under eculizumab therapy are being carried to dissect the key alterations under complement C5 blockade.

The current study is based on use of high-throughput methods to investigate PILs, including exome sequencing (for the non-CHAPLE PILs), transcriptomics, proteome and microbiome investigations. The aims of the study include; 1. Discovery of signatures and biomarkers in CHAPLE, 2. Identification of the molecular etiology of non-CHAPLE PILs and potentially discover novel gene defects. The integrated application of genomics, transcriptome, proteomics and microbiome aims to identify key mediators and pathways operative in the pathogenesis of intestinal lymphangiectasias. Serial evaluation and longitudinal follow up of patient samples under eculizumab (anti-complement C5 antibody) therapy investigates dynamic alterations in the pathological profiles in CHAPLE syndrome. It is anticipiated that these studies will improve the diagnosis and treatment of CHAPLE and related conditions.

Goals of the current study include:

1. To discover novel gene defects underlying PILs not related to CD55 deficiency.
2. To identify signatures of CHAPLE disease and non-CHAPLE PILs that may reveal key mediators of disease and additional novel therapeutic targets.
3. To explore the efficacy of eculizumab in a larger group of CHAPLE patients from unrelated families, with variable degree of disease severity.
4. To analyze patient samples collected before and during eculizumab therapy with the following objectives:

   1. To understand relations between eculizumab concentration, complement function (CH50, AH50) and complement protein levels (C3, C5, CFB, C3a, C5a, sC5b-9, Bb, Ba)
   2. To explore biomarkers of inflammation and thrombosis, complications of the disease that can occur in certain affected individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with PIL form the study groups and deem eligible for the study unless there is a risk associated with blood draw.
2. The patients with CHAPLE syndrome who receive eculizumab therapy and consent to participate in this study are followed prospectively and clinical data collected. Biological sample collection and molecular investigations are to be made only if the patient is willing to provide biological samples, including peripheral blood and stool.

Exclusion Criteria:

1. Presence of a concomitant disease that leads to hypoproteinemia at the time of starting eculizumab such as a urinary protein loss or a hepatic disease that affects production of proteins by liver.
2. A concomitant disease that leads to secondary intestinal lymphangiectasia such as a fontan procedure for congenital heart disease.
3. Unstable clinical condition not allowing blood draw, such as severe anemia.

Max Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All PIL patients, including CHAPLE and non-CHAPLE PILs are to be included in the study.Among the CHAPLE patients who receive eculizumab therapy a prospective follow-up is made. Age matched healthy subjects form the control group.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Reversal of protein-losing enteropathy | 3-6 months
  Serum levels of blood proteins should be normalized. At least 2 out of 3 parameters including albumin, total protein and immunoglobulin G should reach age-specific normal range.
Reversal of patient-specific major symptoms | 12-18 months
  The major symptoms are variable in CHAPLE patients. The symptoms present in a particular patient should be corrected under therapy.

SECONDARY OUTCOMES:
Reversal of other systemic components of the disease. | 12-18 months
  E.g., thrombosis, enterocolitis, micronutrient deficiency, etc.
Correction of previous biochemical and radiological abnormalities | 6-18 months
  E.g., micronutrient deficiency, thrombocytosis; bowell wall thickening, contrast enhancement, recanalization of a thrombotic vessel segment, etc.
Cessation of previous medications | 3-18 months
  Continueed need for previous medications to treat various manifestations of CHAPLE syndrome will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Lenardo, M.D., Study Director — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozen A. CHAPLE syndrome uncovers the primary role of complement in a familial form of Waldmann's disease. Immunol Rev. 2019 Jan;287(1):20-32. doi: 10.1111/imr.12715. PMID 30565236
- [Background] Ozen A, Comrie WA, Lenardo MJ. CD55 Deficiency and Protein-Losing Enteropathy. N Engl J Med. 2017 Oct 12;377(15):1499-1500. doi: 10.1056/NEJMc1710011. No abstract available. PMID 29020581
- [Background] Ozen A, Comrie WA, Ardy RC, Dominguez Conde C, Dalgic B, Beser OF, Morawski AR, Karakoc-Aydiner E, Tutar E, Baris S, Ozcay F, Serwas NK, Zhang Y, Matthews HF, Pittaluga S, Folio LR, Unlusoy Aksu A, McElwee JJ, Krolo A, Kiykim A, Baris Z, Gulsan M, Ogulur I, Snapper SB, Houwen RHJ, Leavis HL, Ertem D, Kain R, Sari S, Erkan T, Su HC, Boztug K, Lenardo MJ. CD55 Deficiency, Early-Onset Protein-Losing Enteropathy, and Thrombosis. N Engl J Med. 2017 Jul 6;377(1):52-61. doi: 10.1056/NEJMoa1615887. Epub 2017 Jun 28. PMID 28657829
- [Background] Kurolap A, Eshach Adiv O, Hershkovitz T, Tabib A, Karbian N, Paperna T, Mory A, Vachyan A, Slijper N, Steinberg R, Zohar Y, Mevorach D, Baris Feldman H. Eculizumab Is Safe and Effective as a Long-term Treatment for Protein-losing Enteropathy Due to CD55 Deficiency. J Pediatr Gastroenterol Nutr. 2019 Mar;68(3):325-333. doi: 10.1097/MPG.0000000000002198. PMID 30418410
- [Background] Kurolap A, Eshach-Adiv O, Hershkovitz T, Paperna T, Mory A, Oz-Levi D, Zohar Y, Mandel H, Chezar J, Azoulay D, Peleg S, Half EE, Yahalom V, Finkel L, Weissbrod O, Geiger D, Tabib A, Shaoul R, Magen D, Bonstein L, Mevorach D, Baris HN. Loss of CD55 in Eculizumab-Responsive Protein-Losing Enteropathy. N Engl J Med. 2017 Jul 6;377(1):87-89. doi: 10.1056/NEJMc1707173. Epub 2017 Jun 28. No abstract available. PMID 28657861